CLINICAL TRIAL: NCT00377650
Title: Polish-Italian-Hungarian RAndomized ThrombEctomy Trial. PIHRATE Trial.
Brief Title: Polish-Italian-Hungarian RAndomized ThrombEctomy Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jagiellonian University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JagiellonianU
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Last update posted 2007-01-17 (Estimated); Status verified 2007-01

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Thrombectomy

INTERVENTIONS:
Device: Percutaneous thrombectomy

SUMMARY:
Aim Primary percutaneous coronary intervention efficacy improvement by DIVER CE thrombectomy system leading to thrombus reduction.

Study design:

Multicenter, prospective, opened, randomized.

Primary endpoints:

ST resolution >70% 60 minutes after PCI

Secondary endpoints:

Thrombectomy system efficacy/passing trough lesion with thrombus reduction according do TIMI thrombus scale ≥ 1 TIMI 3 flow after PCI MBG 3 CMR - infarct size, measurement of left ventricular end-diastolic EDV and end-systolic volumes ESV and ejection fraction (EF) ECHO: measurement of left ventricular end-diastolic EDV and end-systolic volumes ESV, ejection fraction (EF) and wall motion score index (WMSI) Major cardiac events /cardiac death, reMI, rePCI (TVR, TLR, non infarct involved vessel) or CABG/ 6 month follow up Rate of composite angiographic adverse events including: distal embolisation, transient no-reflow or slow flow, final TIMI <3, need of bail out GpIIb/IIIa inhibitors or adenosine or nitroprosside, final thrombus score >1

ELIGIBILITY:
Inclusion Criteria:

* ST elevation acute myocardial infarction within 6 hours since pain onset, with 2 mm ST segment elevation in two lead
* Minimum 3 mm ST segment elevation in one leads
* Vessel reference diameter > 2.5 mm
* When vessel reference diameter ≥ 4,0 mm than additional distal protection device (filter) is needed during stent implantation

Exclusion Criteria:

* Contraindications to PCI (contrast allergy, no possibility to stent implantation) ASA, thienopirydins or GP IIb/IIIa inhibitors
* Active bleeding or coagutopathy
* Prior CABG or PCI
* Known ejection fraction EF <35%
* Cardiogenic shock /SBP < 90 mmHg, IABP and/or catheloamins usage/
* LBBB, pacemaker rhythm
* Severe calcifications
* Previous Myocardial infarction
* Stroke history
* Patient directly after reanimation
* Known thrombocytopenia- platelets < 100 000
* Pregnancy
* Cancer disease
* No future patient cooperation expected
* Patient's taking part in the other clinical trials
* Fibrynolisis directly administered before PCI
* Renal insufficiency (creatynine > 220 µmol/ml), hemodialysis
* Contraindications to PCI (contrast allergy, no possibility to stent implantation) ASA, thienopirydins or GP IIb/IIIa inhibitors
* Active bleeding or coagutopathy
* Prior CABG or PCI
* Known ejection fraction EF <35%
* Cardiogenic shock /SBP < 90 mmHg, IABP and/or catheloamins usage/
* LBBB, pacemaker rhythm
* Severe calcifications
* Previous Myocardial infarction
* Stroke history
* Patient directly after reanimation
* Known thrombocytopenia- platelets < 100 000
* Pregnancy
* Cancer disease
* No future patient cooperation expected
* Patient's taking part in the other clinical trials
* Fibrynolisis directly administered before PCI
* Renal insufficiency (creatynine > 220 µmol/ml), hemodialysis
* Liver insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-09; Study Completion 2007-12

PRIMARY OUTCOMES:
ST resolution >70% 60 minutes after PCI

SECONDARY OUTCOMES:
Thrombectomy system efficacy/passing trough lesion with thrombus reduction according do TIMI thrombus scale ≥ 1
TIMI 3 flow after PCI
MBG 3
CMR - infarct size, measurement of left ventricular end-diastolic EDV and end-systolic volumes ESV and ejection fraction (EF)
ECHO: measurement of left ventricular end-diastolic EDV and end-systolic volumes ESV, ejection fraction (EF) and wall motion score index (WMSI)
Major cardiac events /cardiac death, reMI, rePCI (TVR, TLR, non infarct involved vessel) or CABG/ 6 month follow up
Rate of composite angiographic adverse events including: distal embolisation, transient no-reflow or slow flow, final TIMI <3, need of bail out GpIIb/IIIa inhibitors or adenosine or nitroprosside, final thrombus score >1

CONTACTS AND LOCATIONS:
Overall Officials: Dariusz Dudek, MD, Principal Investigator — Jagiellonian University
Locations (9):
- Institute, Medical School of University Pecs, Pécs, Hungary
- Italy (2):
  - Cardiology Department Hospital Villascassi, Genova
  - Institute of Cardiology, Catholic University, Rome
- Poland (6):
  - Górnośląskie Centrum Medyczne, Katowice
  - Zaklad Hemodynamiki i Angiokardiohrafii IK CMUJ, Krakow
  - Oddział Kardiologii Inwazyjnej, Elektroterapii i Angiologii NZOZ, Nowy Sącz
  - Szpital Wojewódzki w Przemyślu, Przemyśl
  - Instytut Kardiologii im.Prymasa Tysiaclecia Sefana Kardynala Wyszynskiego, Warsaw
  - Slaskie Centrum Chorob Serca, Zabrze

REFERENCES:
- [Derived] Dudek D, Mielecki W, Burzotta F, Gasior M, Witkowski A, Horvath IG, Legutko J, Ochala A, Rubartelli P, Wojdyla RM, Siudak Z, Buchta P, Pregowski J, Aradi D, Machnik A, Hawranek M, Rakowski T, Dziewierz A, Zmudka K. Thrombus aspiration followed by direct stenting: a novel strategy of primary percutaneous coronary intervention in ST-segment elevation myocardial infarction. Results of the Polish-Italian-Hungarian RAndomized ThrombEctomy Trial (PIHRATE Trial). Am Heart J. 2010 Nov;160(5):966-72. doi: 10.1016/j.ahj.2010.07.024. PMID 21095287